CLINICAL TRIAL: NCT06703151
Title: The Benefits of Improving Self-care Ability for Farmers and Fishermen With Existing Cardiometabolic Diseases
Brief Title: To Understand the Self-care Ability of Farmers and Fishermen With CMDs (Hypertension, Heart Disease, Hyperlipidemia, Type 2 Diabetes), Whether They Are Aware of CMDs, Their Treatment Status, Treatment Effectiveness, and Their Ability to Describe Known and Practice the Self-care Content of CMDs.
Acronym: CMDs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Mei-Yen, Chen, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 202301844B0; MOST 113-2314-B-255-002-MY3 (Other Grant/Funding Number: National Science and Technology Council)
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Disease; Diabetes; Hyperlipidemia; Stroke
Keywords: board game; sustainable development goals; climate change; reduced inequalities; cardiometabolic diseases; agriculture; aquaculture; self-care; dehydration status; inflammatory biomarkers
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Hyperlipidemias; Stroke

STUDY DESIGN:
Intervention Model Description: The 1st year will involve a cross-sectional descriptive study targeting farmers and fishermen in the southwest coastal regions. Collaborating with the local health bureau and regional hospitals. It will investigate their self-care abilities, chronic dehydration, and associated influencing factors. The estimated samples are approximately 338 individuals. The research methods for the 2nd and 3rd years involve: (1) Developing a tabletop game educational tool tailored to the socioeconomic and cultural needs of farmers and fishermen, and training designated educators; (2) Employing a community-based quasi-experimental research design. Eligible participants will be cluster-randomized into intervention and control groups. Both groups will receive educational materials. The intervention group will additionally engage with the [SC-8 Monopoly-style board game] intervention, while the control group will only follow the regular community care model.
Masking Description: Structured and semi-structured questionnaires:
  Basic social demographics and health history: age, gender, education level, occupational profile, living status, height, weight, and whether there are chronic diseases diagnosed by a physician, stroke, cancer or immune system-related diseases, etc., current treatment status (treatment method, home implementation overview, treatment institution), how effective the treatment is (biochemical indicators: such as blood pressure, blood sugar, blood lipids); whether there are professionals from medical institutions Provide health information related to personal diseases, such as drug precautions (time, dosage, usage), basic simple home instrument measurements (such as blood pressure monitors, blood glucose machines, weight scales), and self-care related information obtained by patients from medical institutions, weight loss methods and other information (such as diet, calories, exercise, drugs).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group will have (CMDs self-care) teaching material and a [Monopoly board game] plan (Experimental): 1st-5th month: Complete the assessment of self-care ability and biochemical indicators, introduce the (CMDs self-care) teaching material manual, and evaluate the case's referral treatment status from the institution, and provide answers to questions. Played the Monopoly board game 8 times: On average, each community has about 2-3 groups (a group of 4-7 people), each group has a leader (seed teacher) to provide CMDs health education Q&A before each board game activity . The 6th month: Conduct self-care process assessment in each community. The 7th-12th month: Telephone visits are provided every 2 months (3 times in total), each case lasts 5-10 minutes each time.
  Interventions: Behavioral: CMDs (Cardiometabolic Diseases) Self-Care Manual
- Only follow the community screening abnormality handling process and accept the referral treatment (No Intervention): After completing the assessment of self-care ability and biochemical indicators, use the referral treatment and care model of the health center or cooperative hospital; provide self-care manuals to each community in the first to second months, and providing answers to questions (same as the experimental group); conduct self-care process assessments in each community in the 24th week

INTERVENTIONS:
Behavioral: CMDs (Cardiometabolic Diseases) Self-Care Manual — 1st-5th month: Complete the assessment of self-care ability and biochemical indicators, introduce the (CMDs self-care) teaching material manual, and evaluate the case's referral treatment status from the institution, and provide answers to questions. Played the Monopoly board game 8 times: On average, each community has about 2-3 groups (a group of 4-7 people), each group has a leader (seed teacher) to conduct CMDs health education Q&A before each board game activity . 6th month: Conduct self-care process assessment in each community. 7th-12th month: Telephone visits are provided every 2 months (3 times in total), each case lasts 5-10 minutes each time.
  Arms: The experimental group will have (CMDs self-care) teaching material and a [Monopoly board game] plan

SUMMARY:
This project will be based on nursing scholar Dorothea Orem's self-care theory, integrating the concept of the [life essential 8, LE8] proposed by the American Heart Association, as well as our team's recent research findings. We aim to develop educational materials and tools tailored for this group, termed [Self-Care Eight Essentials] aligning with these theories and previous research outcomes. This study aims to present an overview of self-care abilities among farmers and fishermen with cardiovascular and metabolic diseases, identifying the distance from the ideal level and related influencing factors. It intends to establish self-care educational materials and tools tailored to the socioeconomic background of this specific population. Additionally, the study aims to transform these materials into tabletop game educational tools that possess credibility, effectiveness, and an element of entertainment. Through patents and technology transfer, these tools are expected to serve as convenient and effective guidance instruments for health bureaus and primary healthcare units.

DETAILED DESCRIPTION:
Research background: In addition to emphasizing three-stage and five-level prevention strategies, community nursing is also expected to demonstrate innovative capabilities and initiatives in health equality and climate change response in sustainable development. Agriculture and aquaculture are an important development of the country, the foundation of people's life and ecological conservation; Taiwan's southwestern coast is an important base for providing high-quality agricultural and fishery products to the people, accounting for one-third of the households and people engaged in agriculture and fishery in the country. However, with international economic and trade pressures and climate change, the number of these farmers and fishermen is decreasing year by year as they face declining production capacity and income. According to the preliminary research results of our team, the prevalence and mortality rate of cardiometabolic diseases among farmers and fishermen along the southwestern coast are higher than those in the country and advanced countries in Europe and the United States. At the same time, the rate of chronic dehydration is also high. Overall farmers and fishermen have low education levels, are aging, and lack medical resources. Relatively inadequate. Literature shows that if people with cardiometabolic diseases improve their self-care abilities, they can avoid health deterioration such as myocardial infarction and stroke. From the perspective of assisting the sustainable development of agriculture and fisheries, how to overcome the health inequalities caused by social factors determining health? Through The focus of this project is to provide innovative strategies that are consistent with their socio-economic background and to effectively improve their self-care abilities and chronic dehydration problems. In the past, our team has gradually reduced the incidence of liver cancer and other related cancers in the region through the detection, referral and treatment of type C virus hepatitis with a high prevalence in the region. It has also provided the Ministry of Agriculture with relevant health needs and policy initiatives for farmers and fishermen, and has gained a lot of popularity. The trust and attention of relevant units will help us continue to promote cross-domain cooperation. So far, there is a lack of relevant literature at home and abroad to explore and improve the health problems of farmers and fishermen; there is even less research on community nursing to prevent and improve the worsening of cardiometabolic diseases.

Research purpose: Therefore, this project will be based on the results of previous research to conduct the following discussions: (1) the self-care ability of farmers and fishermen with cardiometabolic diseases; (2) designing a design that is consistent with the socio-economic background of farmers and fishermen to improve their self-care Ability teaching materials and teaching aids; (3) Verify the effectiveness of this teaching materials, teaching aids and the experimental design of this study, as a basis for industry-university cooperation with local governments and private enterprises, in order to achieve the influence of benefit diffusion.

Research methods and objects: This project will be based on the self-care theory of nursing scholar Dorothea Orem, combined with the concept of the eight key elements of life [life essential 8, LE8] proposed by the American Heart Association, and the research results of our team in recent years, to construct a structure that is suitable for this group Teaching materials and teaching aids for [Self-care - Octathlon]. This project is expected to be completed in three years. In the first year, a cross-sectional descriptive research method will be used to target farmers and fishermen on the southwest coast. It will cooperate with the Health Bureau and regional hospitals to identify farmers and fishermen with existing cardiometabolic diseases and carry out self-care. To discuss ability, chronic dehydration and its influencing factors, the sample size is estimated to be approximately 338 people. The research methods and purposes in the second to third years are: (1) Complete [board game] teaching aids that meet the socio-economic and cultural background needs of farmers and fishermen, and train seed teachers; (2) Community-based quasi-experimental research design, select Participants in the conditions were randomly assigned to the intervention group and the control group in clusters. Participants in both groups received the [Self-Care-8thlon-SC-8] teaching materials; the intervention group also received the [SC-8-Monopoly Board Game] program. After adopting the conventional community care model with the control group, the differences in self-care ability, cardiometabolic and inflammatory indicators are estimated to be approximately 205 in both groups at this stage. Use descriptive and inferential statistical analysis, such as chi-square and variance tests, multivariable linear, logistic regression and generalized estimating equations, to process repeated measurement data and adjust the effects of influencing factors.

Analysis: The study will employ both descriptive and inferential statistical analyses, such as chi-square and analysis of variance (ANOVA), multivariate linear regression, logistic regression, and generalized estimating equations (GEE) to handle repeated measures data and adjust for the effects of influencing factors.

Expected results: This study will be able to present an overview of the self-care ability of farmers and fishermen with cardiovascular and metabolic diseases, as well as the distance from ideal and related influencing factors, establish self-care teaching materials and teaching aids suitable for the socio-economic background of this group, and transform it into a reliable Through the completion of patents and technology transfer, the [board game] teaching aids with validity and entertaining functions are expected to be used as convenient and effective guidance tools for health bureaus and primary medical care units.

ELIGIBILITY:
Inclusion Criteria:

* Farmers and fishermen who have been diagnosed with CMDs
* Aged between 18 and 75 years old
* Able to take care of their own daily life and can walk to the unit or community activity center that cooperates with this project
* Can communicate with Taiwanese and Mandarin, and agree to participate in the second and third years of this study

Exclusion Criteria:

* Those who have no household registration or live in an unstable place in the study area
* Those who have had a stroke or myocardial infarction
* Those who have kidney and heart failure diseases and have limited water intake
* Those who have cognitive or mental disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The Number of participants who can reduce cardiometabolic risks through enhancing CMDs self-care ability | 12 months
  Conducting CMDs' self-care health education intervention to evaluate participants' health-related behaviour changes and cardiometabolic risks reduction

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Yen Chen, Distinguished Professor, Principal Investigator — Chang Gung University of Science and Technology
Locations (1):
- Chang Gung Memorial Hospital, Mailiao, Yun Lin Hsien, Taiwan

IPD SHARING:
Plan to Share IPD: No
Before share IPD, we want to wait until this study is actually implemented and has concreted physical results.

REFERENCES:
- See also: Report on rural household registration sampling survey in Taiwan — https://www.afa.gov.tw/cht/index.php?act=download&ids=28395
- See also: Ministry of Health and Welfare.Guidelines for preventive care of cardiovascular disease. — https://www.hpa.gov.tw/Pages/EBook.aspx?nodeid=4609
- See also: Health Promotion Administration. Metabolic syndrome. — https://www.hpa.gov.tw/Pages/List.aspx?nodeid=359
- See also: United Nations (2023). Transforming our world: the 2030 agenda for sustainable development goals. — https://sdgs.un.org/goals
- See also: WHO guideline on self-care interventions for health and well-being. — https://www.who.int/publications/i/item/9789240052192

DOCUMENTS (1):
  • Study Protocol (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT06703151/Prot_000.pdf